CLINICAL TRIAL: NCT02063308
Title: Oxaloacetate Pharmacokinetics and Safety
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Russell Swerdlow, MD (Other)
Responsible Party: Sponsor-Investigator, Russell Swerdlow, MD, Gene and Marge Sweeney Professor of Neurology, University of Kansas Medical Center
Organization: University of Kansas Medical Center (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: STUDY00000581
Record Dates: First submitted 2014-02-12; First posted 2014-02-14 (Estimated); Last update posted 2014-07-24 (Estimated); Status verified 2014-07

CONDITIONS: Alzheimer's Disease
Keywords: Oxaloacetate; OAA; AD; Alzheimer's Disease
MeSH Terms: conditions — Alzheimer Disease | interventions — Oxaloacetic Acid

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Oxaloacetate (OAA) (Experimental): 100 mg OAA to be taken twice daily over the course of a month
  Interventions: Dietary Supplement: Oxaloacetate (OAA)

INTERVENTIONS:
Dietary Supplement: Oxaloacetate (OAA)

SUMMARY:
By doing this study, researchers hope to learn how much oxaloacetate (OAA) ends up in the blood after OAA capsules are swallowed, and to assess whether persons with Alzheimer's disease who take OAA for one month have any side-effects.

ELIGIBILITY:
Inclusion Criteria:

* Meet criteria for Mild or Moderate AD
* Have a study partner
* Speak English as primary language.

Exclusion Criteria:

* Absence of a study partner
* Report a potentially confounding, serious medical risk such as type 1 diabetes, cancer, or a recent cardiac event (i.e. heart attack, angioplasty, etc.)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 6 (Actual)
Dates: Start 2014-02; Primary Completion 2014-06 (Actual); Study Completion 2014-06 (Actual)

PRIMARY OUTCOMES:
Correlation between oral OAA intake and plasma levels | Change from dose to 30, 45, 60, 75, 90, 105, 120, 135, 150, and 240 minutes after dosing
  Baseline blood sample will be obtained before 100 mg OAA is administered. Blood samples to be drawn every 15 minutes starting 30 minutes after OAA administration.

SECONDARY OUTCOMES:
safety of OAA in study participants | Change from Baseline to Month 1
  We will evaluate weights, blood counts, electrolytes, liver function tests, insulin levels, and plasma amino acid levels in subjects exposed to OAA for 1 month. These multiple measures will be used to generate a composite safety outcome measure.

CONTACTS AND LOCATIONS:
Overall Officials: Russell Swerdlow, MD, Principal Investigator — University of Kansas Medical Center
Locations (1):
- University of Kansas Medical Center, Kansas City, Kansas, United States